CLINICAL TRIAL: NCT05461664
Title: Avapritinib in the Treatment of Unresectable or Recurrent Metastatic Gastrointestinal Stromal Tumors Non-exon18 Mutations of PDGFRA:A Real-world Study
Brief Title: Avapritinib in the Treatment of Unresectable or Recurrent Metastatic GIST Non-exon18 Mutations of PDGFRA
Status: Recruiting | Type: Observational
Sponsor: Xinhua Zhang, MD (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Fudan University (Other); Peking University People's Hospital (Other); Chinese PLA General Hospital (Other); Xiangya Hospital of Central South University (Other); Peking University Shenzhen Hospital (Other); Nanfang Hospital, Southern Medical University (Other); West China Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Shanghai Zhongshan Hospital (Other); Sun Yat-sen University (Other); Xijing Hospital (Other); Shengjing Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other); Liaoning Cancer Hospital & Institute (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Fujian Medical University Union Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); First Affiliated Hospital of Chongqing Medical University (Other); Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Xinhua Zhang, MD, First Affiliated Hospital, Sun Yat-Sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: No.[2022]107
Record Dates: First submitted 2022-07-09; First posted 2022-07-18 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Gastrointestinal Stromal Tumors; Unresectable Solid Tumor; Recurrent Metastatic Malignant Neoplasm
Keywords: Avapritinib; Genetic testing
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, multicenter, observational real-world study to explore the Avapritinib therapy in GIST patients who definited Non-exon18 Mutations of PDGFRA.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE Gastrointestinal stromal tumors (GIST) are thought to develop from the interstitial cells of Cajal or their stem cell precursors. They are the most common mesenchymal tumors occurring in the gastrointestinal (GI) tract. The annual incidence of GIST is about 1/100,000 ~ 2/100,000 globally. Biological behavior can range from benign to malignant, and immunohistochemical staining is usually positive for CDs 117 and DOG-1, showing Cajal cell differentiation. Eighty-five percent of GISTs is caused by activating mutations in the receptor tyrosine kinase KIT or platelet-derived growth factor receptor alpha (PDGFRA) gene. Targeted therapy for KIT and PDGFRA alters metastatic or unresectable GISTs without effective drug therapy, allowing tumor control and significantly prolonging patient survival.

Following the marketing application approved in March 2021 for Avapritinib and Repaitinib (the indication for the former is GIST with PDGFRA exon18 mutation and the latter is the standard four-line therapy for GIST), five targeted drugs are currently available for treatment of unresectable or recurrent metastatic GIST. The first, second and third-line treatments were imatinib, sunitinib and regorafenib, respectively. Different targeting drugs can inhibit the activation of GIST- or PDGFRA--encoded transmembrane tyrosine kinases by binding to GIST- driven genes to induce apoptosis. There were differences in molecular structure and mechanism of action among the five targeted drugs, which led to different mutations in different exons of GIST, and the sensitivity to targeted drugs was different. KIT protein is a common type III receptor tyrosine kinase (RTK), which is a transmembrane receptor protein. PDGFRA protein is highly homologous and has similar functions. KIT proteins are predominantly extracellular (encoded by exon 9), transmembrane, near-membrane (encoded by exon 11), kinase domains (further divided into kinase binding domains encoded by exon 13/14, and activation loops encoded by exon 17/18). KIT protein has two kinds of three-dimensional spatial conformation (type I-activated conformation and type II-non-activated conformation), which can be transformed and dynamically balanced under normal conditions. The first-line targeted drug imatinib can competitively bind to ATP in the kinase-binding domain of RTK, and the mechanism of action of imatinib is that after the ATP-binding site of the kinase domain is occupied by it, it blocks substrate phosphorylation and signal transduction, inhibits the proliferation of tumor cells and promotes apoptosis. More than 80% of all GISTs in the advanced stage of treatment present as KIT single-gene driven types, and therefore, the clinical benefit rate of first-line imatinib is more than 84%. One of the reasons for primary resistance to first-line therapy is that tumors derive from primary mutations in the activated loop, such as PDGFRA exon 18 D842V mutations, which cause the kinase to tend to an activated conformation for most of the time, whereas imatinib, sunitinib, and regorafenib belong to the same type II TKIs (tyrosine kinase inhibitors), which theoretically can only bind to kinase in a non-activated conformation and are therefore primary resistant to this mutant GIST. In addition, secondary resistance occurs after first-line treatment is effective, with a median of PFS 24 months. The most common cause of resistance is mutations in the KIT gene at the secondary site. The most common secondary mutations are almost concentrated in the exon 13/14 and exon 17/18 regions. Mutations encoding binding domains (exon 13 and 14) prevented the binding of imatinib to RTKs; Mutations that encode activated rings (exon 17 and 18) cause KIT to tend to activate the conformation, preventing most TKIs, including imatinib, from binding to it. Avapritinib is the only type I TKI that has been approved for the treatment of GIST compared to the other 4 targeted agents. Previous studies have found that this compound has a strong inhibitory effect on KIT exon17 D816V mutants that cause mast cell hyperplasia. The mutant is located in the activation ring. Mutations that are highly similar in structure and function are multidrug resistant PDGFRA exon18 D842V mutations accounting for around GIST 5%. Preclinical studies showed broad-spectrum inhibition of KIT or PDGFRA, including KIT exon 11,17,18, and PDGFRA exon 18 mutations, weak affinity for wild-type KIT and PDGFRA, PDGFRB, CSF1R, and FLT3. In the Phase 1 clinical study in patients with metastatic or unresectable PDGFRA D842V-mutant GISTs, the objective response rate (ORR) for Avapritinib was 91%, with a complete response rate of 13%, median duration of efficacy (DOR) of 27.6 m (95% CI 17.6-N%), and median progression-free survival (PFS) of 34 m (95% CI 22.9-N%), with an estimated overall survival (OS) of 61% at 36months. In patients with KIT or non-D842V PDGFRA mutations treated more than three lines, atorvastatin ORRs were 17%, all in partial response (PRs), median DORs were 10.2 m (95% CI 7.% -10.2), clinical benefit rate (CBRs) were 38%, median PFSs were 3.7 m (95% CI 2.% -4.6), and median OSs were 11.6 m (95% CI 9.% -12.6). These studies indicate that Avapritinib is effective in PDGFRA exon 18, especially in the D842V mutant GISTs, and that some of the remaining KIT mutations can also be treated with Avapritinib for tumor control. In vitro studies suggest that KIT activating ring mutations GISTs are sensitive to Avapritinib, but there are no clinical studies evaluating the exact efficacy of Avapritinib in this type of patient population. In addition, on the surface of the preliminary study, secondary resistance to the PDGFRA exon 18 mutation GIST following the benefit of Avapritinib was due to secondary mutations in the PDGFRA gene; However, the causes of secondary resistance to KIT-mutant GISTs that have been shown to be effective in the treatment of Avapritinib and changes in the driver gene are unknown.

Therefore, it is necessary to conduct a multicenter observational study in patients with unresectable or relapsed/metastatic GISTs other than PDGFRA exon 18 mutations in order to explore the benefit of Avapritinib in addition to PDGFRA exon 18 mutations, and to investigate changes in the status of primary and secondary resistance mutations of Avapritinib in order to provide evidence for individualized treatment of advanced GISTs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged ≥ 18 years.
* Gastrointestinal stromal tumors confirmed by histopathological examination, and CD- and/or DOG-1-positive by immunohistochemistry.
* Presence of mRECIST v1.1-compliant lesions with at least one measurable lesion (non-lymphadenopathy ≥1.0 cm or ≥2-fold scan slice thickness).
* Treatment with Avapritinib.
* Patients with an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2 at screening.
* Patient informed consent and signed written consent form.
* The patient was compliant and voluntarily scheduled for follow-up, treatment, laboratory tests, and other study procedures.

Exclusion Criteria:

* KIT or PDGFRA wild type.
* Failure to complete continuous atorvastatin for at least 15 days due to intolerability or disease progression.
* Other serious acute or chronic physical or mental problems, or laboratory abnormalities, may increase the risk associated with participation in the study or use of drugs, or interfere with the judgment of the study results and, in the judgment of the investigator, are not considered appropriate for participation in the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 74 patients with metastatic or unresectable advanced gastrointestinal stromal tumors from tier-3 hospitals who meet the criteria will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  To evaluate objective response rate (ORR,CR+PR) determined by radiology assessment per mRECIST(Response Evaluation Criteriain Solid Tumours), version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.
Clinical Benefit Rate | 2 years
  To evaluate clinical benefit rate(CBR,CR+PR+>16 weeks continuation SD) determined by radiology assessment per mRECIST, version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.
Duration Of Response | 2 years
  To evaluate duration of response (DOR) determined by radiology assessment per mRECIST, version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.If a lesion reappears after disappearing in a patient with complete response, progressive disease is declared. However, if such a lesion behaves in this manner in a patient with stable disease or partial response, it is the change in sum of target disease that defines the response or progression.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  To evaluate PFS determined by radiology assessment per mRECIST, version 1.1 in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.If a lesion reappears after disappearing in a patient with complete response, progressive disease is declared. However, if such a lesion behaves in this manner in a patient with stable disease or partial response, it is the change in sum of target disease that defines the response or progression.
overall survival | 2 years
  To evaluate OS determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
  To evaluate OS determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.Complete response is the disappearance of all lesions with nodes measuring < 10 mm and normal tumour markers.A decrease in the sum of target disease of ≥ 30% represents partial response.Stable disease lies between partial response and progressive disease.If a lesion reappears after disappearing in a patient with complete response, progressive disease is declared. However, if such a lesion behaves in this manner in a patient with stable disease or partial response, it is the change in sum of target disease that defines the response or progression.
Treatment-emergent adverse events | 2 years
  To evaluate treatment-emergent adverse events determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
adverse events of special interest | 2 years
  To evaluate adverse events of special interest determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.
serious adverse events | 2 years
  To evaluate serious adverse events determined in patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Zhang, PhD, Principal Investigator — First affiliated hosptial,Sun Yat-sen university
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Background] Fletcher CD, Berman JJ, Corless C, Gorstein F, Lasota J, Longley BJ, Miettinen M, O'Leary TJ, Remotti H, Rubin BP, Shmookler B, Sobin LH, Weiss SW. Diagnosis of gastrointestinal stromal tumors: A consensus approach. Hum Pathol. 2002 May;33(5):459-65. doi: 10.1053/hupa.2002.123545. PMID 12094370
- [Background] von Mehren M, Joensuu H. Gastrointestinal Stromal Tumors. J Clin Oncol. 2018 Jan 10;36(2):136-143. doi: 10.1200/JCO.2017.74.9705. Epub 2017 Dec 8. PMID 29220298
- [Background] 中国临床肿瘤学会胃肠间质瘤专家委员会. 中国胃肠间质瘤诊断治疗共识（2017 年版）. 肿瘤综合治疗电子杂志. 2018;4(1): 31-42.
- [Background] Ducimetiere F, Lurkin A, Ranchere-Vince D, Decouvelaere AV, Peoc'h M, Istier L, Chalabreysse P, Muller C, Alberti L, Bringuier PP, Scoazec JY, Schott AM, Bergeron C, Cellier D, Blay JY, Ray-Coquard I. Incidence of sarcoma histotypes and molecular subtypes in a prospective epidemiological study with central pathology review and molecular testing. PLoS One. 2011;6(8):e20294. doi: 10.1371/journal.pone.0020294. Epub 2011 Aug 3. PMID 21826194
- [Background] Heinrich MC, Corless CL, Demetri GD, Blanke CD, von Mehren M, Joensuu H, McGreevey LS, Chen CJ, Van den Abbeele AD, Druker BJ, Kiese B, Eisenberg B, Roberts PJ, Singer S, Fletcher CD, Silberman S, Dimitrijevic S, Fletcher JA. Kinase mutations and imatinib response in patients with metastatic gastrointestinal stromal tumor. J Clin Oncol. 2003 Dec 1;21(23):4342-9. doi: 10.1200/JCO.2003.04.190. PMID 14645423
- [Background] Scheijen B, Griffin JD. Tyrosine kinase oncogenes in normal hematopoiesis and hematological disease. Oncogene. 2002 May 13;21(21):3314-33. doi: 10.1038/sj.onc.1205317. PMID 12032772
- [Background] Debiec-Rychter M, Sciot R, Le Cesne A, Schlemmer M, Hohenberger P, van Oosterom AT, Blay JY, Leyvraz S, Stul M, Casali PG, Zalcberg J, Verweij J, Van Glabbeke M, Hagemeijer A, Judson I; EORTC Soft Tissue and Bone Sarcoma Group; Italian Sarcoma Group; Australasian GastroIntestinal Trials Group. KIT mutations and dose selection for imatinib in patients with advanced gastrointestinal stromal tumours. Eur J Cancer. 2006 May;42(8):1093-103. doi: 10.1016/j.ejca.2006.01.030. Epub 2006 Apr 18. PMID 16624552
- [Background] Evans EK, Gardino AK, Kim JL, Hodous BL, Shutes A, Davis A, Zhu XJ, Schmidt-Kittler O, Wilson D, Wilson K, DiPietro L, Zhang Y, Brooijmans N, LaBranche TP, Wozniak A, Gebreyohannes YK, Schoffski P, Heinrich MC, DeAngelo DJ, Miller S, Wolf B, Kohl N, Guzi T, Lydon N, Boral A, Lengauer C. A precision therapy against cancers driven by KIT/PDGFRA mutations. Sci Transl Med. 2017 Nov 1;9(414):eaao1690. doi: 10.1126/scitranslmed.aao1690. PMID 29093181
- [Background] Gebreyohannes YK, Wozniak A, Zhai ME, Wellens J, Cornillie J, Vanleeuw U, Evans E, Gardino AK, Lengauer C, Debiec-Rychter M, Sciot R, Schoffski P. Robust Activity of Avapritinib, Potent and Highly Selective Inhibitor of Mutated KIT, in Patient-derived Xenograft Models of Gastrointestinal Stromal Tumors. Clin Cancer Res. 2019 Jan 15;25(2):609-618. doi: 10.1158/1078-0432.CCR-18-1858. Epub 2018 Oct 1. PMID 30274985
- [Background] Heinrich MC, Jones RL, von Mehren M, Schoffski P, Serrano C, Kang YK, Cassier PA, Mir O, Eskens F, Tap WD, Rutkowski P, Chawla SP, Trent J, Tugnait M, Evans EK, Lauz T, Zhou T, Roche M, Wolf BB, Bauer S, George S. Avapritinib in advanced PDGFRA D842V-mutant gastrointestinal stromal tumour (NAVIGATOR): a multicentre, open-label, phase 1 trial. Lancet Oncol. 2020 Jul;21(7):935-946. doi: 10.1016/S1470-2045(20)30269-2. PMID 32615108
- [Background] Jones RL, Serrano C, von Mehren M, George S, Heinrich MC, Kang YK, Schoffski P, Cassier PA, Mir O, Chawla SP, Eskens FALM, Rutkowski P, Tap WD, Zhou T, Roche M, Bauer S. Avapritinib in unresectable or metastatic PDGFRA D842V-mutant gastrointestinal stromal tumours: Long-term efficacy and safety data from the NAVIGATOR phase I trial. Eur J Cancer. 2021 Mar;145:132-142. doi: 10.1016/j.ejca.2020.12.008. Epub 2021 Jan 16. PMID 33465704
- [Background] George S, Jones RL, Bauer S, Kang YK, Schoffski P, Eskens F, Mir O, Cassier PA, Serrano C, Tap WD, Trent J, Rutkowski P, Patel S, Chawla SP, Meiri E, Gordon M, Zhou T, Roche M, Heinrich MC, von Mehren M. Avapritinib in Patients With Advanced Gastrointestinal Stromal Tumors Following at Least Three Prior Lines of Therapy. Oncologist. 2021 Apr;26(4):e639-e649. doi: 10.1002/onco.13674. Epub 2021 Feb 1. PMID 33453089
- [Background] Grunewald S, Klug LR, Muhlenberg T, Lategahn J, Falkenhorst J, Town A, Ehrt C, Wardelmann E, Hartmann W, Schildhaus HU, Treckmann J, Fletcher JA, Jung S, Czodrowski P, Miller S, Schmidt-Kittler O, Rauh D, Heinrich MC, Bauer S. Resistance to Avapritinib in PDGFRA-Driven GIST Is Caused by Secondary Mutations in the PDGFRA Kinase Domain. Cancer Discov. 2021 Jan;11(1):108-125. doi: 10.1158/2159-8290.CD-20-0487. Epub 2020 Sep 24. PMID 32972961